CLINICAL TRIAL: NCT01673958
Title: The Effect of Stair Descending and Stair Ascending Exercise on Muscle Strength and Performance: the SmartEscalator Device
Brief Title: Stair Descending vs. Stair Ascending Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Collaborators: University of Thessaly (Other); Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dr. Anastasios Theodorou, Principal investigator, European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EUC-011
Record Dates: First submitted 2012-08-22; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Aging; Heart Failure; Sarcopenia
Keywords: Eccentric exercise; Aging; Heart failure; Muscle strength loss; Sarcopenia
MeSH Terms: conditions — Heart Failure; Sarcopenia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stair descending group (Experimental): Stair descending exercise. Participants will carry out six weeks of stair descending training consisting of three exercise sessions per week.
  Interventions: Other: Exercise
- Stair ascending group (Experimental): Stair ascending exercise. Participants will carry out six weeks of stair descending training consisting of three exercise sessions per week.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Comparison between stair descending and stair ascending training

SUMMARY:
The aim of the present project is to compare the acute and chronic effect of stair descending versus stair ascending exercise on muscle damage and performance in elderly males with chronic heart failure.

DETAILED DESCRIPTION:
Study design:

Twelve elderly males with chronic heart failure, New York Heart Association class I-II, will participate in this study. Participants will be allocated into two equally-sized groups: a stair descending group (n = 6) and a stair ascending group (n = 6). At the beginning of the study, the volunteers will perform an acute bout of stair descending or stair ascending exercise on an automatic escalator (4 sets of 3 min each, speed will be set at 45 steps∙min-1). Step height will be 20.5 mm. Before and at day 2 post exercise, physiologic measurements will be performed and blood samples will be collected. Then, participants will carry out six weeks of stair descending or ascending training consisting of three exercise sessions per week (the first two weeks the speed will be set at 45 steps∙min-1, the next two weeks at 50 steps∙min-1 and the last two weeks at 55 steps∙min-1 for both groups). Afterward, they will repeat the acute stair descending or ascending protocol, as carried out at the beginning of the study, and the same physiologic measurements will be performed and blood samples will be collected.

Measurements:

Isometric (at 90 knee flexion), concentric and eccentric peak torque at 60o∙s-1of quadriceps femoris, pain-free range of motion, delayed onset muscle soreness and creatine kinase will be measured.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure (New York Heart Association class I-II)
* subject provides written informed consent
* personal physician of the participants provides written informed consent

Exclusion Criteria:

* smoker
* consumed any nutritional supplement the last 3 months
* performed intense eccentric exercise the last 6 months
* non Caucasian

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Muscle strength (torque) | Change from baseline in muscle strength at day 2 post exercise at the first and sixth week of training
  An isokinetic dynamometer (Cybex, Ronkonkoma, NY) will be used for the measurement of isometric, eccentric and concentric knee extensor peak torque at 90° knee flexion. The average of the three best maximal voluntary contractions with their dominant leg will be recorded. In order to ensure that the subjects provide their maximal effort, the measurements will be repeated if the difference between the lower and the higher torque value exceeded 10%. There will be two minutes rest between isometric efforts.

SECONDARY OUTCOMES:
Pain free range of motion (degrees) | Before and at day 2 post exercise at the first and sixth week of training
  The assessment of pain-free ROM will be performed manually using the the isokinetic dynamometer. The investigator will move the calf at a very low angular velocity from 0 knee extension to the position where the subject will feel any discomfort.
Creatine kinase, CK (activity IU) | Before and at day 2 post exercise at the first and sixth week of training
  CK activity will be measured as a general indicator of muscle damage.It will be measured in a Cobas Integra Plus 400 chemistry analyzer.
Delayed onset muscle soreness, DOMS (scale 1-10) | Before and at day 2 post exercise at the first and sixth week of training
  Each participant will assess delayed onset muscle soreness (DOMS) during squat movement (90o knee flexion) and perceived soreness will be rated on a scale ranging from 1 (normal) to 10 (very sore).

CONTACTS AND LOCATIONS:
Overall Officials: George Panayiotou, PhD, Study Chair — Research Centre, European University Cyprus
Locations (1):
- European University Cyprus, Nicosia, Cyprus

REFERENCES:
- [Background] Paschalis V, Nikolaidis MG, Theodorou AA, Panayiotou G, Fatouros IG, Koutedakis Y, Jamurtas AZ. A weekly bout of eccentric exercise is sufficient to induce health-promoting effects. Med Sci Sports Exerc. 2011 Jan;43(1):64-73. doi: 10.1249/MSS.0b013e3181e91d90. PMID 20508540